CLINICAL TRIAL: NCT02379689
Title: A Randomized, Double-Blinded, Placebo-Controlled With Crossover Study to Evaluate the Efficacy of Intradiscal Injection of Viable Placental Tissue Extract in Subjects With One or Two Level, Symptomatic Lumbar Intervertebral Disc Degeneration
Brief Title: Efficacy of Intradiscal Injection of Viable Placental Tissue Extract in Subjects With One or Two Level, Symptomatic Lumbar Intervertebral Disc Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmes-Murphey Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Parker 1001
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Degenerative Disc Disease; Pain
Keywords: psychosocial state
MeSH Terms: conditions — Intervertebral Disc Degeneration; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- injectable placental tissue extract called BioDGenesis (Active Comparator): This study will compare injectable placental tissue extract called BioDGenesis (Active Product)
  Interventions: Drug: Injectable placental tissue extract called BioDGenesis (Active Product)
- Placebo (Placebo Comparator): injectable Tissue Suspension Solution (TSS) (Placebo). The Active Product is supplied by BioD, LLC (BioD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Injectable placental tissue extract called BioDGenesis (Active Product)
  Arms: injectable placental tissue extract called BioDGenesis
Drug: Placebo
  Arms: Placebo

SUMMARY:
Dr. Parker (the "Investigator") and Semmes Murphey Foundation ("Foundation") are conducting a study of outcomes and safety associated with degenerative discs at Semmes-Murphey Clinic, P.C. ("Semmes-Murphey"). This study will look at a product that is derived from human tissue, that will be injected into the affected disc. With this study, the investigators hope to find a safe and effective way to treat degenerative disc disease.

DETAILED DESCRIPTION:
Dr. Parker (the "Investigator") and Semmes Murphey Foundation ("Foundation") are conducting a study of outcomes and safety associated with degenerative discs at Semmes-Murphey Clinic, P.C. ("Semmes-Murphey"). This study will look at a product that is derived from human tissue, that will be injected into the affected disc. With this study, we hope to find a safe and effective way to treat degenerative disc disease.

This study will compare injectable placental tissue extract called BioDGenesis ("Active Product") to injectable Normal Saline ("Placebo"). The Active Product is supplied by BioD, LLC ("BioD"). You have a 50 percent chance of receiving the Placebo

The study will last for 52 weeks. After all patients have been enrolled in the study and have completed 26 weeks, the Investigator will conduct a safety and efficacy analysis. If the investigator determines that the Active Product is more effective than Placebo in treating degenerative disc disease and there are no safety concerns with the Active Product, patients who received Placebo will have the option of receiving the Active Product through week 52.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be ≥18 and ≤75 years of age, skeletally mature, and have a BMI ≥18 kg/m2 and ≤30 kg/m2 at Screening.
2. The subject must have been experiencing low back pain for at least 6 months prior to Screening.
3. The subject must have had low back pain that is unresponsive to at least 3 months of conservative care (non operative treatment), which may include bed rest, anti inflammatory or analgesic medications, chiropractic manipulations, acupuncture, massage, physical therapy or home-directed lumbar exercise programs.
4. The subject must have pretreatment (Baseline) low back pain of 30 to 90 mm on the visual analog scale (VAS) at Screening and Baseline.
5. The subject must have pretreatment (Baseline) Oswestry Disability Index Questionnaire (ODI) score of 30 to 70 points at Screening and Baseline.
6. The subject's target disc must meet the following objective criteria (corresponding to Pfirrman Grade 2 and 3):
7. The subject must be willing to voluntarily sign the informed consent form and agree to the release of medical information for purposes of this study (i.e., HIPAA authorization) at Screening.
8. The subject must be physically and mentally able to comply with the protocol, able to read and complete the required forms, and willing and able to adhere to the requirements of the protocol.

Exclusion Criteria:

1. The subject has radiculopathy resulting from nerve compression at Screening or Baseline.
2. The subject has unilateral or bilateral leg pain with intensity greater than 50% of the intensity of the low back pain as measured on a VAS at Screening or Baseline.
3. The subject has cauda equina syndrome at Screening or Baseline (Day 1).
4. The subject has greater than 50% loss of disc height when compared to the adjacent superior disc.
5. The subject has a significant disc herniation or free fragment of disc material on MRI.
6. The subject has current infection at the planned procedure site, active systemic infection, or current or prior history of lumbar spinal infection (i.e., discitis, septic arthritis, epidural abscess) at Baseline.
7. The subject has had previous lumbar spine surgery.
8. The subject has had previous disc treatment procedures or intradiscal injections. Discography may have been performed, but the procedure must have been done at least 2 weeks or more prior to the injection of study medication.
9. The subject has undergone lumbar epidural or transforaminal injections with corticosteroids within the last 3 months.
10. The subject has evidence of prior lumbar vertebral body fracture or trauma.
11. The subject has evidence of dynamic instability on lumbar flexion extension.
12. The subject has Grade 2 or higher spondylolisthesis or spondylolysis at the target disc at Screening.
13. The subject has findings of a significant underlying neurological condition (motor strength <4; sensory assessment abnormal; or reflexes absent or hyperactive with clonus).
14. The subject has an active malignancy or tumor.
15. The subject has had significant systemic disease, such as unstable angina, autoimmune disease, rheumatoid arthritis, diabetes mellitus, or muscular dystrophy.
16. The subject has a coagulopathy or thrombocytopenia.
17. The subject is currently taking anticoagulant, antineoplastic, antiplatelet, or thrombocytopenia inducing medications (except for aspirin or nonsteroidal anti-inflammatory drugs [NSAIDS]) at Baseline.
18. The subject is taking opioid analgesics regularly more than 2 times per day, or taking long acting or long term opioids for more than 90 days at Baseline.
19. The subject has concomitant conditions requiring daily oral steroid usage for more than 30 days in the preceding 90 days before Screening.
20. The subject has a history of unexplained, easy, or persistent bruising or bleeding, bleeding from the gums, or bleeding problems experienced in previous surgical procedures.
21. The subject has a history of hypersensitivity or anaphylactic reaction to bovine products, HA, or dimethyl sulfoxide (DMSO).
22. The subject is currently using tobacco or has actively used tobacco within 3 months prior to enrollment.
23. The subject has an uncontrolled psychiatric condition or substance/alcohol abuse that would potentially interfere with the subject's participation in the study within 2 years prior to Screening.
24. The subject has participated in another drug or device clinical study within the 2 months immediately prior to Screening.
25. The subject is known to be pregnant or nursing at time of enrollment or with plans to become pregnant within the planned length of the study.
26. The subject has pending litigation against a health care professional or other pending civil litigation, except where required by the insurer as a condition of coverage.
27. The subject has active or pending worker's compensation claims.
28. The subject has a body habitus that precludes adequate fluoroscopic visualization for the procedure or the procedure is physically impossible.
29. The subject has a contraindication to MRI scanning or cannot tolerate MRI scanning.

    -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
• To evaluate the effect on change from baseline compared to Tissue Suspension Solution of intradiscal placental extract (IPE) on lower back pain (VAS). | 52 weeks
• To evaluate the effect on change from baseline compared to Tissue Suspension Solution of intradiscal placental extract on disability (ODI). | 52 weeks
• To evaluate the effect on change from baseline compared to Tissue Suspension Solution of intradiscal placental extract on quality of life (EQ-5D). | 52 weeks

SECONDARY OUTCOMES:
• Composite outcome measure: Change from baseline and compared to Tissue Suspension Solution in qualitative assessments | 52 weeks
  • Composite outcome measure: Change from baseline and compared to Tissue Suspension Solution in qualitative assessments associated with MRI imaging (T2-weighted image), including Pfirrman score, modic changes, annular tears/fissures, endplate integrity, herniation and additional observations at 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Institutional Review Board® (WIRB®), Puyallup, Washington, Washington, United States